CLINICAL TRIAL: NCT03768596
Title: Nudging for Vaccination : Efficacity and Acceptability Among Medical Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adriaan Barbaroux (Individual)
Collaborators: Université de Nice Sophia Antipolis (Other)
Responsible Party: Sponsor-Investigator, Adriaan Barbaroux, Principal Investigator, Barbaroux, Adriaan, M.D.
Organization: Barbaroux, Adriaan, M.D. (Individual)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ABarbaroux; 2018-A02939-46 (Other: ID RCB)
Record Dates: First submitted 2018-12-05; First posted 2018-12-07 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Influenza, Human; Vaccination; Sepsis
Keywords: Nudge; acceptability
MeSH Terms: conditions — Influenza, Human; Sepsis

STUDY DESIGN:
Intervention Model Description: one group receives a form with the nudge, one group receives the same form without nudge and another group doesn't receive any form
Masking Description: In the first pat of the study, participants are unaware of the fact we are trying to nudge them. In the second part, they are explained and asked what they feel about nudging
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nudge (Experimental): receiving nudge and form
  Interventions: Behavioral: Nudge; Other: vaccination form
- No nudge (Active Comparator): receiving the same form without nudge (only questions about their opinion/attitudes about vaccination)
  Interventions: Other: vaccination form
- No intervention (No Intervention): receiving no nudge nor form

INTERVENTIONS:
Behavioral: Nudge — Influenza Vaccine Prescription Form accompanied on the back of telephone numbers of occupational health centers of different hospitals where interns are likely to be on probation.
  Arms: Nudge
Other: vaccination form — a form about vaccination
  Arms: No nudge; Nudge

SUMMARY:
Nudge is a set of methods aimed at helping people adopt a behavior by a gentle prompt, conscious or not. Classically, Nudges rely on heuristics and cognitive biases. These methods have been studied for years in social psychology and are receiving renewed attention since the awarding of the Nobel Prize in economics to Richard Thaler for his work on the application of Nudge to the economy.

Health professionals are very inadequately vaccinated (25 to 45% of the population). Some studies have shown that a Nudge based on intent implementation can significantly increase vaccination coverage. However, few studies evaluate the acceptability of Nudge or its application to health professionals.

The investigators sought to apply a Nudge based on availability heuristics to health professionals, in order to evaluate its effectiveness and terms of behavior adoption (influenza vaccination) and its acceptability.

The investigator's hypothesis is that Nudging is both effective and acceptable and that people found nudging more acceptable if they have been exposed to a nudge.

DETAILED DESCRIPTION:
The investigators asked residents in general medicine to pass a questionnaire including a Nudge. This Nudge was the influenza vaccine prescription form accompanied on the back of the telephone numbers of the occupational health centers of the hospitals where residents were on probation.

The interns of the group "Nudge" saw at the end of their questionnaire the following statement: "If you are not vaccinated against the flu so far, you can get the form stapled to this questionnaire, it will allow you to get the vaccine in pharmacy. On the back you will also find practical information about immunization services at your place of training. " A group will receive an implemented Nudge questionnaire, a group will receive a questionnaire without Nudge and a control group will not be asked. (Phase 1) The 3 groups will receive a month later a questionnaire evaluating the effectiveness in terms of immunization coverage, and the acceptability of the Nudge, for oneself and for others. (Phase 2) The control group will only receive the Phase 2 questionnaire to control the Hawthorne effect.

The difference between the 3 groups will consist exclusively in the exposure of the participants to:

* A questionnaire on their attitude (opinion) towards vaccination;
* The numbers of the occupational health vaccination centers of their places of training;
* The flu vaccine prescription form, to be signed and stamped by a doctor (also already freely available on the internet)

ELIGIBILITY:
Inclusion Criteria:

* medical students

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Efficiency: vaccination rate | 1 month
  vaccination rate

SECONDARY OUTCOMES:
acceptability: scale | One month
  likert based acceptability form

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle MILHABET, MD, PhD, Study Chair — LAPCOS-UCA
Locations (1):
- UNSA, Nice, France

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: starting 6 months after publication
Access Criteria: OK for meta analysis, please contact directly Dr Adriaan BARBAROUX.

REFERENCES:
- [Derived] Barbaroux A, Benoit L, Raymondie RA, Milhabet I. Nudging health care workers towards a flu shot: reminders are accepted but not necessarily effective. A randomized controlled study among residents in general practice in France. Fam Pract. 2021 Jul 28;38(4):410-415. doi: 10.1093/fampra/cmab001. PMID 33506858